CLINICAL TRIAL: NCT00820950
Title: A Double-Blind, Vehicle-Controlled, Rising Dose, Safety, Tolerability, Pharmacokinetic and Preliminary Efficacy Study of Ruxolitinib Phosphate Cream When Applied to Patients With Plaque Psoriasis
Brief Title: A Study of Ruxolitinib Phosphate Cream When Applied to Patients With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-201
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort A: INCB018424 Ruxolitinib 0.5% (Experimental): INCB018424 Ruxolitinib 0.5% vs vehicle applied once daily for 28 days
  Interventions: Drug: Ruxolitinib phosphate cream; Drug: Placebo cream
- Cohort B: INCB018424 Ruxolitinib 1.0% (Experimental): INCB018424 Ruxolitinib 1.0% vs vehicle applied once daily for 28 days
  Interventions: Drug: Placebo cream; Drug: Ruxolitinib phosphate cream
- Cohort C: INCB018424 Ruxolitinib 1.5% (Experimental): INCB018424 Ruxolitinib 1.5% vs vehicle applied twice for 28 days
  Interventions: Drug: Placebo cream; Drug: Ruxolitinib phosphate cream
- Cohort D: 18424 Ruxolitinib vs Dovonex® calcipotriene (Experimental): INCB018424 up to 1.5% versus Dovonex® calcipotriene 0.005% cream applied BID for 28 days
  Interventions: Drug: Dovonex® calcipotriene 0.005%
- Cohort E: 18424 Ruxolitinib vs Diprolene® AF betamethasone diproprionate (Experimental): INCB018424 up to 1.5% versus Diprolene ® AF betamethasone dipropionate 0.05% cream applied twice a day for 28 days
  Interventions: Drug: Diprolene® AF betamethasone dipropionate 0.05% cream.

INTERVENTIONS:
Drug: Ruxolitinib phosphate cream — Ruxolitinib phosphate cream 0.5%
  Other Names: INCB018424
  Arms: Cohort A: INCB018424 Ruxolitinib 0.5%
Drug: Dovonex® calcipotriene 0.005% — Cream applied once or twice daily for up to 56 days.
  Arms: Cohort D: 18424 Ruxolitinib vs Dovonex® calcipotriene
Drug: Diprolene® AF betamethasone dipropionate 0.05% cream. — Cream applied once or twice daily for up to 56 days
  Arms: Cohort E: 18424 Ruxolitinib vs Diprolene® AF betamethasone diproprionate
Drug: Placebo cream — Cream applied once or twice daily for 56 days
  Arms: Cohort A: INCB018424 Ruxolitinib 0.5%; Cohort B: INCB018424 Ruxolitinib 1.0%; Cohort C: INCB018424 Ruxolitinib 1.5%
Drug: Ruxolitinib phosphate cream — Ruxolitinib phosphate cream 1.0%
  Other Names: INCB018424
  Arms: Cohort B: INCB018424 Ruxolitinib 1.0%
Drug: Ruxolitinib phosphate cream — Ruxolitinib phosphate cream 1.5%
  Other Names: INCB018424
  Arms: Cohort C: INCB018424 Ruxolitinib 1.5%

SUMMARY:
The study is comprised of two parts. The first portion of this study will be a double-blind, Sponsor-unblinded, vehicle-controlled study with application of ruxolitinib or vehicle to paired lesions at least 15 cm apart in patients with active but stable plaque psoriasis. Part 2 of the study is a double-blind, sponsor unblinded, comparison of ruxolitinib with two FDA approved products in patients with active but stable plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 17 to 40 kg/m2
* Subjects must have two comparable psoriatic lesions measuring between 9 and 100 cm2 and these target lesions must be similar in size to each other, and separated by at least 15 cm.

Exclusion Criteria:

* Subjects with lesions solely involving the palms of the hands or soles of the feet or intertriginous areas, the scalp or the face.
* Subjects with pustular psoriasis or erythroderma.
* Subjects currently on other topical agents or UVB therapy within 2 weeks of the first dose of study medication.
* Subjects receiving PUVA within 4 weeks of the first dose of study medication.
* Subjects receiving systemic retinoids, etanercept, adalimumab or efalizumab or oral immunosuppressives within 3 months prior to the first dose of study medication.
* Subjects receiving any other biological therapy (infliximab, alefacept, abatacept, etc) within 3 months of the first dose of study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-05-31 (Actual); Primary Completion 2009-01-31 (Actual); Study Completion 2009-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Williams, MD, Study Director — Incyte Corporation
Locations (6):
- United States (6):
  - Vallejo, California
  - Boston, Massachusetts
  - Rochester, New York
  - Stony Brook, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Punwani N, Scherle P, Flores R, Shi J, Liang J, Yeleswaram S, Levy R, Williams W, Gottlieb A. Preliminary clinical activity of a topical JAK1/2 inhibitor in the treatment of psoriasis. J Am Acad Dermatol. 2012 Oct;67(4):658-64. doi: 10.1016/j.jaad.2011.12.018. Epub 2012 Jan 24. PMID 22281165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 study centers in the United States from 08 May 2007 to 28 April 2008. This study is completed.
Pre-assignment Details: A total of 29 participants with active but stable plaque psoriasis were enrolled in the 2 part dose escalation study; 27 participant completed the study. In Part 1, each participant treated 1 plaque with INCB018424 cream, and a matching plaque with vehicle cream. In Part 2, each participant treated 1 plaque with INCB018424 cream, and a matching plaque with a comparator drug cream.
Units Other Than Participants: Plaques
Groups:
- Part 1 Cohort A: Vehicle Cream; Part 1 Cohort B: Vehicle Cream; Part 1 Cohort C: Vehicle Cream: Vehicle cream was applied once a day for 28 days
- Part 1 Cohort A Ruxolitinib 0.5% Cream: Ruxolitinib 0.5% was applied once a day for 28 days
- Part 1 Cohort B Ruxolitinib 1.0% Cream: Ruxolitinib 1.0% was applied once a day for 28 days
- Part 1 Cohort C Ruxolitinib 1.5% Cream: Ruxolitinib 1.5% was applied once a day for 28 days
- Part 2 Cohort D: INCB18424: up to 1/5% Ruolitinib cream was applied twice a day for 28 days
- Part 2 Cohort D Calcipotriene (Dovonex®): Calcipotriene (Dovonex®) 0.005% cream was applied twice a day for 28 days
- Part 2 Cohort E: INCB18424: up to 1.5% Ruxolitinib cream was applied twice a day
- Part 2 Cohort E Betamethasone Dipropionate (Diprolene® AF): Betamethasone Dipropionate (Diprolene® AF) 0.05% cream were applied twice a day for 28 days
Period: Overall Study
Arm/Group | Part 1 Cohort A: Vehicle Cream | Part 1 Cohort A Ruxolitinib 0.5% Cream | Part 1 Cohort B: Vehicle Cream | Part 1 Cohort B Ruxolitinib 1.0% Cream | Part 1 Cohort C: Vehicle Cream | Part 1 Cohort C Ruxolitinib 1.5% Cream | Part 2 Cohort D: INCB18424 | Part 2 Cohort D Calcipotriene (Dovonex®) | Part 2 Cohort E: INCB18424 | Part 2 Cohort E Betamethasone Dipropionate (Diprolene® AF)
Started | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 5; 5 Plaques | 5; 5 Plaques
Completed | 5; 5 Plaques | 5; 5 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 6; 6 Plaques | 5; 5 Plaques | 5; 5 Plaques | 5; 5 Plaques | 5; 5 Plaques
Not Completed | 1; 1 Plaques | 1; 1 Plaques | 0; 0 Plaques | 0; 0 Plaques | 0; 0 Plaques | 0; 0 Plaques | 1; 1 Plaques | 1; 1 Plaques | 0; 0 Plaques | 0; 0 Plaques
Not completed — Scheduling Conflict | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT included all enrolled participants who received at least 1 dose of INCB018424 cream.
Groups:
- Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream: Ruxolitinib 0.5% vs. vehicle cream once a day for 28 days
- Part 1 Cohort B: Ruxolitinib 1.0% Cream vs. Vehicle Cream: Ruxolitinib 1.0% cream vs. vehicle cream once a day for 28 days
- Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream: Ruxolitinib 1.5% vs. vehicle cream twice a day for 28 days
- Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®): Ruxolitinib up to 1.5% versus Calcipotriene (Dovonex®) 0.005% cream applied twice a day for 28 days
- Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF): Part 2 INCB018424, up to 1.5% cream versus Betamethasone Dipropionate (Diprolene® AF) 0.05% cream applied twice a day for 28 days
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Part 1 Cohort B: Ruxolitinib 1.0% Cream vs. Vehicle Cream | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (14.25) | 48.8 (10.25) | 55.8 (10.38) | 50.2 (21.13) | 46.2 (10.08) | 48.7 (13.79)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 4 | 5 | 4 | 3 | 4 | 20
  Female | 2 | 1 | 2 | 3 | 1 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  White or Caucasian | 5 | 6 | 5 | 6 | 5 | 27
  Other | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 6 | 5 | 6 | 5 | 4 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Target Lesion Individual Component Scores for Erythema, Scaling and Thickness Compared to Baseline
Description: The investigator assessed the severity of the clinical signs erythema, scaling, and thickness for each test site by using a 5-point scale from 0 (no evidence) to 4.0 (severe).
Time Frame: Baseline, Days 8, 15, 22, 28 and 56
Population: Intent-to-Treat (ITT) population; 1 subject in Cohort A discontinued due to a protocol violation (Day 28 visit was late, because subject was on vacation) and 1 subject in Cohort D discontinued due to other reason (scheduling conflicts).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Part 1 Cohort A: Ruxolitinib 0.5% Cream: Ruxolitinib 0.5% once a day for 28 days
- Part 1 Cohort B: Ruxolitinib 1.0% Cream: Ruxolitinib 1.0% cream once a day for 28 days
- Part 1 Cohort C: Vehicle Cream: Vehicle cream was applied twice a day for 28 days
- Part 1 Cohort C: Ruxolitinib 1.5% Cream: Ruxolitinib 1.5% twice a day for 28 days
- Part 2 Cohort D: INCB18424; Part 2 Cohort E: INCB18424: up to 1.5% Ruxolitinib cream was applied twice a day
- Part 2 Cohort D: Calcipotriene (Dovonex®): Calcipotriene (Dovonex®) 0.005% cream was applied twice a day
- Part 2 Cohort E: Betamethasone Dipropionate (Diprolene® AF): Betamethasone Dipropionate (Diprolene® AF) 0.05% cream was applied twice a day for 28 days
Arm/Group | Part 1 Cohort A: Vehicle Cream | Part 1 Cohort A: Ruxolitinib 0.5% Cream | Part 1 Cohort B: Vehicle Cream | Part 1 Cohort B: Ruxolitinib 1.0% Cream | Part 1 Cohort C: Vehicle Cream | Part 1 Cohort C: Ruxolitinib 1.5% Cream | Part 2 Cohort D: INCB18424 | Part 2 Cohort D: Calcipotriene (Dovonex®) | Part 2 Cohort E: INCB18424 | Part 2 Cohort E: Betamethasone Dipropionate (Diprolene® AF)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
Scores on a scale
  Day 8 - Erythema: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 4 | 4
  Day 8 - Erythema | -0.5 (0.84) | -0.5 (0.55) | -0.8 (0.41) | -1.0 (0.63) | -0.7 (0.82) | -1.2 (0.75) | -1.2 (1.10) | -0.8 (0.84) | -1.0 (0.82) | -1.3 (0.96)
  Day 8 - Scaling | -0.2 (0.41) | -0.2 (0.41) | 0.0 (0.00) | -0.2 (0.41) | -0.7 (0.82) | -1.2 (0.41) | -0.6 (0.89) | -0.6 (0.55) | -0.8 (0.50) | -0.8 (0.50)
  Day 8 - Thickness: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 4 | 4
  Day 8 - Thickness | -0.7 (1.03) | -0.7 (1.03) | -0.2 (0.41) | -0.3 (0.52) | -0.3 (0.52) | -0.8 (0.75) | -0.4 (0.89) | -0.6 (0.55) | -0.5 (0.58) | -0.8 (0.96)
  Day 15 - Erythema: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 15 - Erythema | -0.7 (0.82) | -0.7 (0.82) | -0.8 (0.75) | -1.0 (0.63) | -0.5 (0.84) | -1.2 (0.98) | -1.0 (0.71) | -0.8 (0.45) | -1.0 (1.00) | -1.2 (0.84)
  Day 15 - Scaling: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 15 - Scaling | -0.3 (0.52) | -0.3 (0.52) | -0.2 (0.75) | -0.3 (0.82) | -0.7 (0.82) | -1.0 (0.00) | -0.2 (0.84) | -0.4 (0.55) | -0.8 (0.45) | -1.2 (0.45)
  Day 15 - Thickness: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 15 - Thickness | -0.3 (0.52) | -0.3 (0.52) | -0.2 (0.41) | -0.3 (0.52) | -0.5 (0.55) | -0.8 (0.41) | -0.6 (1.14) | -0.8 (0.84) | -0.6 (1.14) | -0.6 (0.89)
  Day 22 - Erythema: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 22 - Erythema | -0.8 (0.84) | -1.0 (0.71) | -1.0 (0.63) | -1.5 (0.84) | -0.3 (0.82) | -1.2 (0.98) | -1.8 (1.30) | -1.0 (1.00) | -1.4 (0.89) | -1.6 (0.55)
  Day 22 - Scaling: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 22 - Scaling | -0.4 (0.55) | -0.6 (0.55) | -0.5 (0.55) | -0.8 (0.75) | -0.5 (0.84) | -1.2 (0.41) | -0.6 (1.14) | -0.6 (0.89) | -0.8 (0.45) | -1.0 (0.71)
  Day 22 - Thickness: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 22 - Thickness | -0.2 (1.10) | -0.6 (0.89) | -0.3 (0.52) | -0.5 (0.84) | -0.8 (0.75) | -1.2 (0.75) | -1.0 (1.00) | -0.8 (0.45) | -1.0 (0.71) | -0.8 (0.84)
  Day 28 - Erythema: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 28 - Erythema | -0.6 (0.55) | -0.4 (0.55) | -1.2 (0.41) | -1.7 (0.52) | -0.5 (0.55) | -1.0 (0.63) | -1.4 (1.14) | -1.2 (0.84) | -1.2 (0.84) | -1.8 (0.84)
  Day 28 - Scaling: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 28 - Scaling | -0.2 (0.45) | -0.4 (0.55) | -0.7 (0.52) | -1.0 (0.63) | -0.5 (0.55) | -1.2 (0.41) | -0.8 (1.10) | -0.8 (0.84) | -0.8 (0.45) | -1.2 (0.84)
  Day 28 - Thickness: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 28 - Thickness | -0.4 (0.55) | -0.2 (0.45) | -0.3 (0.52) | -1.0 (0.63) | -1.2 (0.75) | -1.5 (0.55) | -1.0 (1.00) | -1.0 (0.00) | -1.0 (0.71) | -1.2 (0.45)
  Day 56/ET - Erythema | -0.5 (1.05) | -0.3 (0.52) | 0.0 (0.63) | -0.2 (0.41) | -0.5 (0.84) | -0.5 (0.84) | -1.0 (0.63) | -1.2 (1.47) | 0.2 (0.84) | -0.6 (0.55)
  Day 56/ET - Scaling | -0.2 (0.41) | -0.2 (0.41) | 0.3 (0.82) | 0.7 (0.82) | -0.7 (0.82) | -0.7 (0.82) | -0.8 (0.75) | -0.7 (1.21) | -0.2 (0.84) | -0.4 (0.89)
  Day 56/ET - Thickness | -0.3 (0.52) | -0.3 (0.52) | 0.0 (0.75) | 0.2 (0.75) | -0.7 (1.03) | -0.8 (0.98) | -1.2 (0.75) | -1.0 (0.63) | 0.0 (0.71) | -0.4 (0.55)

2. Primary Outcome: Change in Target Lesion TOTAL Score (Sum of Erythema + Scaling + Thickness) Compared to Baseline
Description: The total target lesion score was calculated by summing the scores for erythema, scaling, and thickness for that particular target lesion. The investigator assessed the severity of the clinical signs erythema, scaling, and thickness for each test site by using a 5-point scale from 0 (no evidence) to 4.0 (severe).
Time Frame: Baseline, Days 8, 15, 22, 28 and 56
Population: ITT population; 1 subject in Cohort A discontinued due to a protocol violation (Day 28 visit was late, because subject was on vacation) and 1 subject in Cohort D discontinued due to other reason (scheduling conflicts)
Measure: Mean (Standard Deviation); unit: Score on Scale
Groups:
- Part 1 Cohort A: Vehicle; Part 1 Cohort B: Vehicle: placebo cream
- Part 1 Cohort B: Ruxolitinib 1.0% Cream vs. Vehicle Cream: Ruxolitinib 1.0% cream once a day for 28 days
- Part 1 Cohort C: Vehicle Cream: Vehicle Placebo cream
- Part 2 Cohort D: INCB18424: up to 1.5% Ruxolitinib
- Part 2 Cohort E: INCB18424: up to 1.5% Ruxolitinib cream
Arm/Group | Part 1 Cohort A: Vehicle | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Part 1 Cohort B: Vehicle | Part 1 Cohort B: Ruxolitinib 1.0% Cream vs. Vehicle Cream | Part 1 Cohort C: Vehicle Cream | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Part 2 Cohort D: INCB18424 | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Part 2 Cohort E: INCB18424 | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
Score on Scale
  Day 8: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 4 | 4
  Day 8 | -1.3 (1.97) | -1.3 (1.21) | -1.0 (0.63) | -1.7 (1.37) | -1.7 (2.07) | -3.2 (1.72) | -2.4 (2.70) | -2.2 (1.79) | -2.3 (0.96) | -2.8 (1.71)
  Day 15: number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 15 | -1.3 (1.75) | -1.3 (1.75) | -1.3 (2.07) | -2.0 (1.79) | -1.7 (2.07) | -3.0 (1.26) | -2.0 (2.55) | -2.2 (1.79) | -2.4 (2.07) | -3.0 (1.87)
  Day 22: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 22 | -1.4 (1.95) | -2.2 (1.79) | -1.8 (0.98) | -3.0 (2.00) | -1.7 (2.25) | -3.5 (1.76) | -3.6 (3.13) | -2.6 (1.82) | -3.2 (1.64) | -3.4 (1.67)
  Day 28: number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 6 | 5 | 5 | 5 | 5
  Day 28 | -1.2 (1.30) | -1.0 (1.41) | -2.2 (1.17) | -3.8 (1.60) | -2.2 (1.60) | -3.7 (1.37) | -3.4 (2.70) | -3.2 (1.30) | -3.0 (1.58) | -4.2 (1.79)
  Day 56/ET | -1.5 (1.87) | -1.3 (1.21) | 0.5 (1.87) | 0.5 (1.38) | -1.8 (2.23) | -2.0 (2.10) | -3.2 (1.60) | -3.0 (2.90) | 0.0 (2.00) | -1.4 (1.67)

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: A TEAE is any AE either reported for first time or worsening of a pre-existing event after first dose of study drug.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B: Ruxolitinib 1.0% Cream Versus Vehicle: Ruxolitinib 1.0% vs. placebo cream once a day for 28 days
Arm/Group | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Cohort B: Ruxolitinib 1.0% Cream Versus Vehicle | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5
Participants | 6 | 1 | 5 | 4 | 2

4. Primary Outcome: Pharmacokinetics Parameter : Skin Flux of INCB018424
Description: The INCB018424 skin flux was estimated from the overall mean steady-state plasma concentrations for each participant.
Time Frame: Days 8, 15, 22, and 28
Measure: Mean (Standard Deviation); unit: ng/cm^2/h
Groups:
- Part 1 Cohort B: Ruxolitinib 1.0% Cream Versus Vehicle: Ruxolitinib 1.0% vs. placebo cream once a day for 28 days
Arm/Group | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Part 1 Cohort B: Ruxolitinib 1.0% Cream Versus Vehicle | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
ng/cm^2/h | 54.2 (40.8) | 151 (70) | 422 (200) | 363 (215) | 383 (256)

5. Primary Outcome: Pharmacokinetics Parameter : Bioavailability of INCB018424
Description: The INCB018424 bioavailability will be estimated from the overall mean steady-state plasma concentrations for each subject in this study and the estimated systemic clearance of INCB018424 following oral-dose administration in another study. Bioavailability is defined as the proportion of a drug which enters the circulation when introduced into the body and so is able to have an active effect.
Time Frame: Days 8, 15, 22, and 28
Measure: Mean (Standard Deviation); unit: Percentage of dosage
Arm/Group | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Cohort B: Ruxolitinib 1.0% Cream Versus Vehicle | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5
Percentage of dosage | 2.8 (3.2) | 3.0 (1.9) | 3.0 (1.9) | 2.7 (1.1) | 2.7 (2.3)

6. Secondary Outcome: Change in Target Lesion Area Compared to Baseline
Description: Lesion area was estimated on Day 1 and Day 28 using a tracings of the lesion on transparency paper and measurement of the area.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: cm^2
Groups:
- Cohort A: Vehicle; Cohort B: Vehicle; Cohort C: Vehicle: Placebo cream
- Cohort D: INCB18424: Ruxolitinb to 1.5%
- Cohort E: INCB18424: Ruxolitinib up to 1.5%
Arm/Group | Cohort A: Vehicle | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Cohort B: Vehicle | Cohort B: Ruxolitinib 1.0% Cream Versus Vehicle | Cohort C: Vehicle | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Cohort D: INCB18424 | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Cohort E: INCB18424 | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5
cm^2 | 0.35 (4.872) | 1.53 (9.760) | 0.45 (3.775) | -3.18 (8.651) | -4.03 (12.303) | -11.45 (13.851) | -5.22 (6.203) | -2.54 (6.778) | 1.53 (1.624) | -0.48 (5.892)

ADVERSE EVENTS:
Time Frame: Up to approximately 2 months
Description: Adverse Events were reported at the participant level, not the treatment level within each cohort.
Groups:
- Total: Total
Arm/Group | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream | Part 1 Cohort B: Ruxolitinib 1.0% Cream vs. Vehicle Cream | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF) | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/29
Other Adverse Events (participants affected / at risk) | 6/6 | 1/6 | 5/6 | 4/6 | 2/5 | 18/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Cohort A: Ruxolitinib 0.5% Cream vs. Vehicle Cream (N=6) | Part 1 Cohort B: Ruxolitinib 1.0% Cream vs. Vehicle Cream (N=6) | Part 1 Cohort C: Ruxolitinib 1.5% Cream vs. Vehicle Cream (N=6) | Part 2 Cohort D: Ruxolitinib vs. Calcipotriene (Dovonex®) (N=6) | Part 2 Cohort E: Ruxolitinib vs. Betamethasone Dipropionate (Diprolene® AF) (N=5) | Total (N=29)
APPLICATION SITE REACTION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 3 (5)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ELECTROCARDIOGRAM QT INTERVAL ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ELECTROCARDIOGRAM T WAVE ABNORMAL (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
FEELING COLD (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
HAEMATOCRIT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RETICULOCYTE COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
URINE KETONE BODY PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement